CLINICAL TRIAL: NCT05715073
Title: Improving Neuroprotection, Cognitive Function, and Mental Focus With Neurodegradation Countermeasure
Brief Title: Improving Cognition With Neurodegradation Countermeasure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor & Chair, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Pro00123869
Record Dates: First submitted 2023-01-06; First posted 2023-02-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hemodynamics; Caffeine; TeaCrine; Cognitive Change
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: This is a crossover intervention, in which participants will partake in all 3 conditions with at least 96 hours of washout between conditions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind study, participants and those involved in data collection and analysis will not know which arm they have been assigned each visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TeaCrine and caffeine (Experimental): 150mg of Teacrine and 150mg of caffeine
  Interventions: Dietary Supplement: TeaCrine and Caffeine
- Caffeine (Active Comparator): 300mg of caffeine
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): 300mg of cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: TeaCrine and Caffeine — Participants will take Teacrine and caffeine then an hour later perform an intense interval exercise protocol followed by cognitive tests.
  Arms: TeaCrine and caffeine
Dietary Supplement: Caffeine — Participants will take caffeine then an hour later perform an intense interval exercise protocol followed by cognitive tests.
  Arms: Caffeine
Other: Placebo — Participants will take the placebo cellulose pill and than an hour later perform an intense interval exercise protocol followed by cognitive tests.
  Arms: Placebo

SUMMARY:
The goal of this randomized, placebo-controlled, three-condition, double-blind, within-participants crossover clinical trial is to compare caffeine, TeaCrine plus caffeine, and a placebo condition in ROTC or tactical personnel.

The main question it aims to answer is the effect of the condition on measures of cognitive performance, cardio-autonomic, and hemodynamic responses after a physically demanding protocol.

The physiological function will be derived from metrics of heart rate variability, whilst cogntive performance will be evaluated using tasks that assess cognitive domains of executive function, reaction time, and memory.

Participants will report to the lab 4 times, once for familiarization of cognitive measures and then 3 times for their experimental visits. Participants will consume their randomized condition an hour prior to the fatiguing interval exercise protocol. Following they will complete a series of cognitive tasks.

DETAILED DESCRIPTION:
The purpose of this randomized, placebo-controlled, three-condition, double-blind, within-participants crossover clinical trial is to determine and compare the effects of the combination of TeaCrine® and caffeine to a placebo and a caffeine condition on measures of cognitive performance, cardio-autonomic, and hemodynamic responses after a physically demanding protocol. After giving informed consent, 20 ROTC members or tactical personnel will undergo baseline performance testing and familiarization and will then be randomly assigned to order of completion of the placebo (P), caffeine (C) condition, and caffeine + TeaCrine (CT) condition, with each session separated by at least 96 hours. In each condition, Participants will be given the condition pill assigned to them, the pill will be taken orally with water, and will wait 60 minutes. At this time, the Participant will complete a treadmill-based physically fatiguing interval protocol with select cognitive testing during the exercise recovery intervals. Participant measures of mental fatigue will be assessed pre- and post-testing, and following the interval bout participants will perform a series of cognitive tasks. Heart rate variability (HRV) and respiration will be assessed continuously though these tasks and blood pressure will be assessed at baseline, prior to the exercise bout, immediately following the exercise bout, and following the cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Participant is in good health and able to participate in high-intensity exercise.
* Participant is physically active: participating in resistance and/or endurance exercise ≥4 d/wk and ≥150 min/wk for ≥6 mo.
* Participant habitually consumes ≤240 mg caffeine/d (the equivalent of 3 cups of coffee).
* Participants will be asked about dietary supplementation use within the past 6 months.

(If Participant began taking a supplement within the past month, the Participant will be asked to discontinue supplement use followed by a 2-week washout prior to participation. In all other cases, supplement use will be asked to be maintained throughout the study).

Exclusion Criteria:

* Participant currently taking any prescription stimulants (i.e., Adderall, Ritalin, Vyvanse, etc.)
* Participant with any metabolic disorder including known electrolyte abnormalities, diabetes, thyroid disease, adrenal disease or hypogonadism.
* Participant with any inborn error of metabolism.
* Participant with a history of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Participant with sickle cell trait.
* Participant with a personal history of heart disease, high blood pressure (systolic >140 mm Hg & diastolic >90 mm Hg), psychiatric disorders, cancer, benign prostate hypertrophy, gastric ulcer, reflux disease, or any other medical condition deemed exclusionary by the medical staff.
* Participant currently taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive, or anti-coagulant medications.
* Participant who has a known allergy to any of the ingredients in the supplement or the placebo.
* Participant who has migraines.
* Participant with a history of caffeine sensitivity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in blood lactate | On the experimental visit days: Min 0 prior to the exercise protocol, minutes 10, 22, and 30 during the exercise protocol, 5 min after the protocol (min 35), 10 minutes post exercise (min 40)
  Changes in blood lactate across the experimental visit
Changes in Autonomic Nervous System Function (ANS) by linear metrics | On the experimental visit days, this will be measured on a second by second basis from the beginning to the end of the visit (approximately 2 hours)
  To determine if the intervention impacts ANS function by measuring heart rate variability represented by linear time domain metrics.
Changes in Autonomic Nervous System Function (ANS) by nonlinear metrics | On the experimental visit days, this will be measured on a second by second basis from the beginning to the end of the visit (approximately 2 hours)
  To determine if the intervention has an impact on ANS function by measuring heart rate variability represented by nonlinear (ApSaEn) time domain metric.
Changes in Autonomic Nervous System Function (ANS) by frequency domain metrics | On the experimental visit days, this will be measured on a second by second basis from the beginning to the end of the visit (approximately 2 hours)
  To determine if the intervention has an impact on ANS function by measuring heart rate variability represented by frequency domain metrics.
Changes in Inhibitory Control by reaction time (Go/No go) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on inhibitory control by measuring reaction time to Go targets (hits).
Changes in Inhibitory Control by reaction time by errors(Go/No go) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on inhibitory control by measuring errors of commission representing incorrect responses to the target NoGo (false alarm).
Changes in Attention (Go/No go) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the device has an impact on attention by measuring errors of omission to the target Go (misses).
Changes in Inhibitory Control by accuracy scores (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on inhibitory control measured by the accuracy scores (% of correct answers) for compatible-congruent, incompatible-congruent, compatible-incongruent, and incompatible-incongruent Flanker Task trials.
Changes in Inhibitory Control by average response time (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on inhibitory control measured by the average response time to incongruent flanker task trials irrespective of compatible or incompatible rule sets.
Changes in Inhibitory Control by commission errors (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  o determine if the intervention has an impact on inhibitory control measured by the commission errors when an individual fails to respond correctly to a flanker task trial, and commission error runs when an individual fails to respond correctly to multiple successive trials.
Changes in Attention by accuracy (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on attention measured by the accuracy scores for congruent-compatible Flanker task trials.
Changes in Attention by average response time (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on attention measured by the overall average response time (milliseconds) to compatible and incompatible Flanker task trails irrespective of trial congruency.
Changes in Attention by omission errors (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on attention measured by the omission errors when an individual fails to respond to a flanker task trial, and omission error runs when an individual fails to respond to multiple successive trials.
Changes in Cognitive flexibility by accuracy (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on cognitive flexibility by the accuracy scores for incongruent-incompatible Flanker task trials.
Changes in Cognitive flexibility by average response time (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on cognitive flexibility measured by the average response time to incongruent-incompatible flanker task trials.
Changes in Cognitive control by post-error accuracy (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on cognitive control measured by post-error accuracy on Flanker task trials following an error.
Changes in Cognitive control by sequential congruency effect (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine changes in cognitive control measured by sequential congruency effect when lower interference occurs following an incongruent relative to a congruent flanker task trial reflecting a consciously controlled narrowing of attention to the central target.
Changes in Cognitive control by inverse efficiency (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on cognitive control measured by inverse efficiency a metric of a speed-accuracy trade-off for Flanker task trials.
Changes in Attentional Inhibition (Flanker Task) | On the experimental visit days: minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an impact on attentional inhibition measured by congruency interference representing the costs associated with the interference demands associated with incongruent vs congruent flanker task trials.
Changes in Rating of Perceived Exertion | On the experimental visit days: baseline at minute 0, minutes 10, 22, and 30 during the exercise protocol, and 30 minutes after the exercise protocol
  To determine if the intervention has an effect on perceived exertion, measured by Borg's Rating of Perceived Exertion scale from 6 to 20. Higher measures indicate more exertion.
Changes in mood Brunel University Mood Scale (BRUMS). | On the experimental visit days: baseline at minute 0, immediately after completion of the exercise protocol at approximately 90 minutes into the visit, and 30 minutes after the exercise protocol approximately 120 minutes into the visit
  To determine if the intervention has an effect on mental fatigue and mood.
Changes in Object Hit and Avoid | On the experimental visit days: Immediately after and 30 minutes after the completion of the exercise protocol.
  To determine the effects of the intervention on rapid response execution and inhibition during complex continuous task performance.
Changes in Anti-Saccade Task | On the experimental visit days: Immediately after and 30 minutes after the completion of the exercise protocol.
  To determine the effects of the intervention on higher level processes, assessing response inhibition, working memory, and visuospatial attention.
Changes in Modified Trail Making Task | On the experimental visit days: Immediately after and 30 minutes after the completion of the exercise protocol.
  To determine the effects of the intervention on visuomotor processing and executive function.
Changes in 2-Back Task | On the experimental visit days: Immediately after and 30 minutes after the completion of the exercise protocol.
  The determine the effects of the intervention on working memory capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No